CLINICAL TRIAL: NCT02034643
Title: Increase of Tracheal Cuff Pressure During Transesophageal Echocardiography Probe Insertion: Double-lumen Tube Versus Single-lumen Tube
Brief Title: Transesophageal Echocardiography(TEE) Probe Insertion and Tracheal Cuff Pressure
Acronym: TEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YSJeon_Cuff
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-01

CONDITIONS: Intubation, Intratracheal

ARMS (2):
- patients with single-lumen tube (Other): Patients who required intraoperative TEE and single-lumen tube; balloon pressure adjustment before TEE probe insertion
  Interventions: Procedure: balloon pressure adjustment
- patients with double-lumen tube (Other): Patients who required intraoperative TEE and double-lumen tube; balloon pressure adjustment before TEE probe insertion
  Interventions: Procedure: balloon pressure adjustment

INTERVENTIONS:
Procedure: balloon pressure adjustment — Tracheal cuff pressure was adjusted to 18 mmHg (25 cmH2O) before TEE probe insertion

SUMMARY:
Tracheal cuff overinflation is known to reduce tracheal mucosal blood flow and to increase tracheal morbidity. Transesophageal echocardiography (TEE) probe insertion may increase the tracheal cuff pressure. The aim of this study is to evaluate the effect of TEE probe insertion on tracheal cuff pressure and to compare the effects in single-lumen tube and double-lumen tube.

ELIGIBILITY:
Inclusion Criteria:

* adult patients scheduled for elective cardiothoracic surgery
* requiring intraoperative TEE monitoring

Exclusion Criteria:

* patients with tracheal stenosis
* patients with tracheoesophageal fistula
* patients with esophageal surgery
* patients with esophageal varix
* patients with Barrett esophagus
* patients with esophageal hernia
* patients with descending thoracic aorta aneurysm
* patients with dysphagia
* patients with vocal fold palsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Tracheal cuff pressure | 1 min after TEE probe insertion

SECONDARY OUTCOMES:
Tracheal cuff pressure | every min for 5 min after TEE probe insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim TK, Min JJ, Seo JH, Lee YH, Ju JW, Bahk JH, Hong DM, Jeon Y. Increased tracheal cuff pressure during insertion of a transoesophageal echocardiography probe: A prospective, observational study. Eur J Anaesthesiol. 2015 Aug;32(8):549-54. doi: 10.1097/EJA.0000000000000204. PMID 25564781